CLINICAL TRIAL: NCT01468519
Title: Effects of Continuous Subcutaneous Insulin Infusion (CSII) on Erectile Dysfunction in T2DM Patients: A Prospective, Exploratory, Controlled Trial
Brief Title: Exploratory CSII Trial on Erectile Dysfunction in T2DM Patients
Acronym: ECSIITED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jothydev's Diabetes and Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Jothydev Kesavadev, CEO & Director., Jothydev's Diabetes and Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JDC/Pump/020/2011
Record Dates: First submitted 2011-07-02; First posted 2011-11-09 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2; Erectile Dysfunction
Keywords: Diabetes mellitus, type 2; Erectile dysfunction; continuous subcutaneous insulin infusion; CSII; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Erectile Dysfunction; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSII (Experimental): continuous subcutaneous insulin infusion
  Interventions: Drug: Insulin
- MDI (Active Comparator): multiple daily insulin injections
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin via continuous subcutaneous insulin infusion
  Arms: CSII
Drug: Insulin — insulin via multiple daily injections
  Arms: MDI

SUMMARY:
Erectile dysfunction (ED) is a common form of organic sexual dysfunction in males with diabetes, with estimated incidence rates between 35 and 75%. Fifty percent of men with diabetes are afflicted with ED within 10 years of their diagnosis. Long-term poor glycemic control increases the risk ED. Although comparatively costly, advantages of CSII over other modes of insulin delivery include better glycemic control, fewer hypoglycemic episodes, and improved quality of life. In a previously published study, on CSII in T2DM, in our center, 83% of men reported an improvement in sexual function as a secondary endpoint. The current study is planned to further explore this finding.

DETAILED DESCRIPTION:
Background Erectile dysfunction (ED) is a common form of organic sexual dysfunction in males with diabetes, with estimated incidence rates between 35 and 75%. Fifty percent of men with diabetes are afflicted with ED within 10 years of their diagnosis. Long-term poor glycemic control increases the risk ED. Neuropathy is a major contributor to diabetic ED. Other causes of ED in diabetes include vascular disease, metabolic control, nutrition, endocrine disorders, psychogenic factors, and drugs.

Continuous Sub-cutaneous Insulin Infusion The Continuous Subcutaneous Insulin Infusion (CSII) Pump (insulin pump for short) is a pager-sized device which can be connected to the body through an infusion set so as to deliver insulin continuously. It consists of a disposable reservoir for insulin, a disposable infusion set, including a cannula for subcutaneous insertion and a tubing system which connects the insulin reservoir to the cannula. Insulin pump therapy by itself is not a new therapy for diabetes mellitus. It is an alternative delivery mechanism for administration of insulin and is found to be superior to ordinary syringes and insulin pens. Insulin pumps were popularly used in T1DM but nowadays insulin pumps are commonly used in T2DM patients as well.

A guideline for use of insulin pumps in India has been recently published in Diabetes Technology and Therapeutics journal, which included participation from Jothydev's Diabetes Center.

Although comparatively costly, advantages of CSII over other modes of insulin delivery include better glycemic control, fewer hypoglycemic episodes, and improved quality of life. Our own center has reported a significant reduction in HbA1c when subjects in multiple daily insulin switched to CSII.

Relevant Clinical Data In the aforementioned study of CSII in Type 2 diabetes patients in our study, 83% of men reported an improvement in sexual function when queried after 6 months on CSII. The mode of improvement and magnitude of this effect is not known, and needs to be ascertained in prospective trials. The present study proposal is to corroborate the findings, and obtain clarification of effect size.

Potential Benefits & Risks The following improvements can be expected following initiation of insulin pump therapy.

* Improvement in HbA1c
* Reduction in blood sugar fluctuations
* Reduction in major and minor hypoglycemic episodes
* Reduction in total daily dose of insulin
* Improvement in QOL

The following are some risks/disadvantages of using insulin pump therapy

* Cost of pumps and consumables is higher than other modes of insulin delivery
* There is a risk of infection if the cannula is not changed once in every three days.
* Improper use of insulin pump boluses can lead to insulin stacking and low sugars.

Proper patient education and monitoring will be part of the study to overcome the risks of insulin pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male T2DM patients with HbA1c < 9%
* Mild ED to Moderate ED as defined by International Index of Erectile Function (IIEF) questionnaire
* Able and willing to use insulin pumps for at least the duration of the study

Exclusion Criteria:

* Severe dysfunction in IIEF Score or duration of ED more than 3 years
* Heart failure (class II - IV) or unstable cardiovascular disease; poorly controlled blood pressure (systolic > 170 or < 90 mmHg or diastolic > 100 or < 50 mmHg) or orthostatic hypotension
* Medications: Substance abuse, anticancer and steroid therapy
* Sexual dysfunction in partner, lack of stable relationship.
* History of radical prostatectomy or pelvic surgery, significant penile deformities, penile implants, or history of stroke or spinal-cord trauma.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in total International Index of Erectile Function (IIEF) score from baseline to six months | baseline and six months
  IIEF quetionnaire is a standardised and validated 15-item self-evaluation scale that provides pre-post treatment clinic evaluations of erectile function, orgasmic function, sexual desire, satisfaction in sexual intercourse and general satisfaction

SECONDARY OUTCOMES:
Global assessment question on erectile function | baseline and 6 months
  Global assessment question (GAQ), "Has the treatment you have been having improved your erections? (yes/no)."

CONTACTS AND LOCATIONS:
Overall Officials: Jothydev Kesavadev, MD, Principal Investigator — Jothydev's Diabetes & Research Center; Gopika Krishnan, BPHARM, Study Chair — Jothydev's Diabetes & Research Center
Locations (1):
- Jothydev's Diabetes & Research Center, Thiruvananthapuram, Kerala, India

REFERENCES:
- [Background] Kesavadev J, Das AK, Unnikrishnan R 1st, Joshi SR, Ramachandran A, Shamsudeen J, Krishnan G, Jothydev S, Mohan V. Use of insulin pumps in India: suggested guidelines based on experience and cultural differences. Diabetes Technol Ther. 2010 Oct;12(10):823-31. doi: 10.1089/dia.2010.0027. PMID 20807118
- [Result] Kesavadev J, Balakrishnan S, Ahammed S, Jothydev S. Reduction of glycosylated hemoglobin following 6 months of continuous subcutaneous insulin infusion in an Indian population with type 2 diabetes. Diabetes Technol Ther. 2009 Aug;11(8):517-21. doi: 10.1089/dia.2008.0128. PMID 19698065
- [Derived] Kesavadev J, Sadasivan Pillai PB, Shankar A, Warrier RS, Ramachandran L, Jothydev S, Krishnan G. Exploratory CSII Randomized Controlled Trial on Erectile Dysfunction in T2DM Patients (ECSIITED). J Diabetes Sci Technol. 2018 Nov;12(6):1252-1253. doi: 10.1177/1932296818794704. Epub 2018 Aug 29. No abstract available. PMID 30156866